CLINICAL TRIAL: NCT04603183
Title: A Randomized, 2-Arm, Open-Label, Ph-II Study of Abemaciclib Combined With ET w/ or w/o CT With Paclitaxel as 1L in Patients With Unresectable Locally Advanced or Metastatic HR(+)/HER2(-) BC With Aggressive Disease Criteria
Brief Title: ABemaciclib, ET ± paclItaxel in aGgressive HR+/HER2- MBC trIaL
Acronym: ABIGAIL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MedSIR (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MedOPP321; 2020-001648-24 (EudraCT Number)
Record Dates: First submitted 2020-10-07; First posted 2020-10-26 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer Metastatic
MeSH Terms: interventions — abemaciclib; Paclitaxel; Letrozole; Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional Arm (Arm A) (Experimental): Abemaciclib 150 mg orally twice daily (BID) during each 28 day cycle combined with ET (2.5 mg letrozole, orally administered and taken daily during each 28-day cycle, or 500 mg fulvestrant, by intramuscular [IM] administration on Days 1 and 15 (±3 days) of the first treatment cycle and Day 1 of each cycle thereafter.
  Interventions: Drug: Abemaciclib; Drug: Letrozole; Drug: Fulvestrant
- Control Arm (Arm B) (Active Comparator): Paclitaxel 90 mg/m² infused over 1 hour on Days 1, 8, and 15 of the 28 day cycle, with at least a 6-day time span between separated doses.
  Interventions: Drug: Paclitaxel

INTERVENTIONS:
Drug: Abemaciclib — Patients will receive abemaciclib 150 mg orally twice daily (BID) (300 mg daily, administered as six 50 mg tablets) during each 28 day cycle combined with either letrozole or fulvestrant.
  Other Names: Verzenios
  Arms: Interventional Arm (Arm A)
Drug: Paclitaxel — Paclitaxel 90 mg/m² infused over 1 hour on Days 1, 8, and 15 of the 28 day cycle, with at least a 6-day time span between separated doses.
  Other Names: Paclitaxel Teva
  Arms: Control Arm (Arm B)
Drug: Letrozole — Patients will receive 2.5 mg letrozole, orally administered and taken daily during each 28-day cycle combined with abemaciclib.
  Arms: Interventional Arm (Arm A)
Drug: Fulvestrant — Patients will receive 500 mg fulvestrant, by intramuscular [IM] administration on Days 1 and 15 (±3 days) of the first treatment cycle and Day 1 of each cycle thereafter combined with abemaciclib.
  Arms: Interventional Arm (Arm A)

SUMMARY:
This is a multicenter, randomized, 2 arm, open label, phase II study. It is designed to compare the efficacy and safety of abemaciclib combined with ET (letrozole or fulvestrant) versus a short course with induction chemotherapy with paclitaxel followed by maintenance therapy with abemaciclib combined with ET (letrozole or fulvestrant) in patients with previously untreated, unresectable locally advanced, or metastatic HR positive/HER2 negative breast cancer with aggressive disease criteria.

DETAILED DESCRIPTION:
The ABIGAIL study aims to provide consistent evidence that the combination of abemaciclib with ET -consisting of letrozole or fulvestrant-as first-line regimen is non-inferior to the optimal first-line chemotherapy -consisting of weekly paclitaxel-in terms of early ORR after the first 12 weeks of treatment in patients with HR-positive/HER2-negative ABC and at least one feature of aggressive disease associated with poor prognosis.

ELIGIBILITY:
Inclusion criteria

1. Signed informed consent form (ICF) prior to participation in any study-related activities.
2. Male or female patients ≥18 years at the time of signing the ICF.
3. Eastern Cooperative Oncology Group performance status of 0 or 1.
4. Life expectancy of at least 24 weeks.
5. Pre-menopausal, peri-menopausal, and post-menopausal women as defined by any of the following criteria:

   1. Documented bilateral oophorectomy;
   2. Age ≥60 years;
   3. Age <60 years and cessation of regular menses for ≥12 consecutive months with no alternative pathological or physiological cause; and serum estradiol and/or FSH level within the laboratory's reference range for post-menopausal females.
6. Unresectable locally advanced or metastatic breast cancer (MBC) that is not amenable to resection with curative intent.
7. At least one of the following aggressive disease criteria:

   1. Presence of visceral disease;
   2. Either radiological as per RECIST v1.1 or clinical evidence of progressive disease (PD) on or within 36 months of completing adjuvant endocrine therapy (ET);
   3. High histological grade and/or PgR-negative status on primary tumor;
   4. LDH >1.5 × the upper limit of normal (ULN).
8. Histologically confirmed estrogen receptor-positive and/or progesterone receptor (PgR)-positive (with ≥1% positive stained cells according to National Comprehensive Cancer Network and American Society of Clinical Oncology guidelines) and HER2-negative (0 to 1+ by immunohistochemistry or 2+ and negative by in situ hybridization test) breast cancer based on local testing on the most recent analyzed biopsy.
9. Measurable disease as per RECIST v1.1 with at least one site of disease amenable to biopsy. Patients with bone lesions as the only sites of metastatic disease are not eligible, except for patients with identifiable soft tissue components, evaluable by cross sectional imaging techniques such as CT or magnetic resonance imaging (MRI), and that meet the definition of measurability according to RECIST v1.1.

   Note: Previously irradiated lesions can only be considered as measurable disease if disease progression has been unequivocally documented at that site since radiation.
10. Willingness and ability to provide a tumor biopsy from a metastatic site or the primary breast tumor at the time of the inclusion and at the time of treatment progression (if feasible) to perform exploratory studies. If not feasible, patient eligibility should be evaluated by Sponsor's qualified designee.
11. Willingness to provide blood samples for exploratory studies at baseline, after 2 weeks (Cycle [C]1, day [D]15) of study treatment, 4 weeks (C2D1), 12 weeks (at the primary efficacy endpoint, corresponding to C4D1), 4 weeks from the initiation of abemaciclib-containing treatment, and at progression (or study treatment termination prior to starting second-line treatment).
12. Willingness to provide stool samples plus Patient-Reported Food Frequency Questionnaires for exploratory studies at study entry (baseline), 4 weeks after the start of treatment (C2D1), and at time of disease progression. Patients on Arm B will also have a stool sample collected 4 weeks from the initiation of abemaciclib-containing treatment.
13. Patients relapsing on a cyclin-dependent kinase (CDK)4/6 inhibitor-based regimen in the neoadjuvant or adjuvant setting will be suitable for the study if disease progression is confirmed after at least 12 months following CDK 4/6 treatment completion.
14. No prior systemic therapy for unresectable locally advanced or metastatic disease.
15. Radiation therapy for metastatic disease is permitted but the patient must have fully recovered from the acute effects and at least 14 days must have elapsed between the last dose and randomization.

    Note: For limited-field radiotherapy, at least 7 days must have elapsed between the last dose and randomization.
16. Resolution of all acute toxic effects of prior anti-cancer therapy to Grade ≤1 as determined by the NCI-CTCAE v 5.0 (except for Grade ≤2 neuropathy, alopecia, or other toxicities not considered a safety risk for the patient at investigator's discretion) within at least 14 days prior to study Day 1.
17. Adequate hematologic and organ function within 14 days before the first study treatment on Day 1 of Cycle 1, defined by the following:

    1. Hematological: White blood cell count >3.0 × 109/L; Absolute neutrophil count ≥1.5 × 109/L (without granulocyte colony-stimulating factor support within 2 weeks prior to Cycle 1, Day 1); Platelet count ≥100 × 109/L (without transfusion within 2 weeks prior to Cycle 1, Day 1); Hemoglobin >9.0 g/dL (without transfusion within 2 weeks prior to Cycle 1, Day 1).
    2. Hepatic:

    i. Serum albumin ≥ 3 g/dL; ii. Total bilirubin ≤ 1.5 × ULN (≤2 × ULN in the case of Gilbert's disease); iii. Aspartate transaminase and alanine transaminase ≤3.0 × ULN (in the case of liver metastases ≤5 × ULN); iv. Alkaline phosphatase ≤2.5 × ULN (in the case of liver and/or bone metastases ≤ 5 × ULN).

    c. Renal: i. Serum creatinine <1.5 × ULN or creatinine clearance ≥30 mL/min based on Cockcroft-Gault glomerular filtration rate estimation.

    d. Coagulation: i. Partial thromboplastin time (or activated partial thromboplastin time and international normalized ratio ≤1.5×ULN.
18. Women of childbearing potential must have a negative serum pregnancy test at 1 week prior to the start of treatment and a further confirmation test on Day 1 (C1D1) before receiving the first dose, and must agree to remain abstinent (refrain from heterosexual intercourse) or to use a medically acceptable method of contraception during the study and for a variable period of time depending on the treatment received thereafter.
19. Men with female partners of childbearing potential or pregnant female partners, must remain abstinent or use a medically acceptable method of contraception during the treatment period and subsequently depending on treatment received.
20. Able to swallow oral medication.
21. Patients who are reliable, willing to be available for the duration of the study and are willing to follow study procedures.

Exclusion criteria

1. Known hypersensitivity to abemaciclib, letrozole, fulvestrant, paclitaxel, and/or any of their excipients.
2. Are currently receiving an investigational drug in a clinical study or participating in any other type of medical research judged not to be scientifically or medically compatible with this study.

   Note: For patients who stopped receiving an investigational drug in another clinical study, a washout period of 21 days or 5-half-lives (whichever is shorter) must be observed before entering the trial.
3. Formal contraindication to ET defined as visceral crisis and rapidly or symptomatic progressive visceral disease.
4. Known concurrent malignancy or malignancy within 5 years of study enrollment except for carcinoma in situ of the cervix, non-melanoma skin carcinoma, or stage I uterine cancer. For other cancers considered to have a low risk of recurrence, discussion with the medical monitor is required.
5. Known active brain metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable for ≥4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable, and without requirement of steroid treatment for ≥14 days prior to first dose of study treatment.
6. Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the study.
7. Major surgical procedure within 14 days prior to treatment initiation or anticipation of the need for a major surgical procedure during the course of the study other than for diagnosis.

   Note: Placement of central venous access catheter(s) (e.g., port or similar) is not considered a major surgical procedure and is therefore permitted.
8. Active bleeding diathesis venous thrombo-embolism, previous history of bleeding diathesis, or chronic anti-coagulation treatment, or any indications or history of Disseminated Intravascular Coagulation (DIC) or Deep vein thrombosis (DVT).
9. Serious and/or uncontrolled pre-existing medical condition(s) that, in the judgment of the investigator, would preclude participation in this study (for example, interstitial lung disease, severe dyspnea at rest or requiring oxygen therapy, severe renal impairment [e.g., estimated creatinine clearance <30 ml/min], history of major surgical resection involving the stomach or small bowel, or pre-existing Crohn's disease or ulcerative colitis or a pre-existing chronic condition resulting in baseline Grade 2 or higher diarrhea).
10. Current known infection with HIV, hepatitis B virus (HBV), or hepatitis C virus (HCV). Patients with past HBV infection or resolved HBV infection (defined as having a negative hepatitis B surface antibody [HBsAg] test and a positive hepatitis B core antibody [HBcAb] test, accompanied by a negative HBV DNA test) are eligible. Patients positive for HCV antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV RNA.
11. Active bacterial or fungal infection at the time of enrolment (requiring antibiotics or antifungal agents at time of initiating study treatment).
12. History of any of the following conditions: syncope of cardiovascular etiology, ventricular arrhythmia of pathological origin (including, but not limited to, ventricular tachycardia and ventricular fibrillation), or sudden cardiac arrest.
13. Pregnant, breastfeeding, or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through a period of 3 weeks to 2 years after the last dose of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2021-06-02 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
12-week overall response rate (ORR) | 12 weeks
  Complete response (CR) or partial response (PR), during the first 12 weeks of treatment as per blinded independent central review, using Response Evaluation Criteria in Solid Tumors (RECIST) version (v) 1.1.

SECONDARY OUTCOMES:
ORR | Baseline up to 24 months
  The best overall response of CR or PR, as per investigator assessment and per blinded independent central review, using RECIST v 1.1.
Clinical benefit rate (CBR) | Baseline up to 24 months
  An objective response (CR or PR), or stable disease for at least 24 weeks, as per investigator assessment and blinded independent central review using RECIST v 1.1.
12-week progression-free survival (PFS) rate | Baseline up to 12 weeks
  The proportion of patients with disease progression or death from any cause, whichever occurs first during the first 12 weeks from randomization, as per investigator assessment and blinded independent central review using RECIST v 1.1.
PFS | Baseline up to 24 months
  The period of time from randomization to the first occurrence of disease progression or death from any cause, whichever occurs first, as per investigator assessment and blinded independent central review using RECIST v 1.1.
Time to response (TTR) | Baseline up to 24 months
  The time from randomization to time of the first objective tumor response (tumor shrinkage of ≥30%) observed in patients who achieved a CR or PR, as per investigator assessment and blinded independent central review using RECIST v 1.1.
Duration of response (DoR) | Baseline up to 24 months
  The time from the first occurrence of a documented objective response to disease progression or death from any cause, whichever occurs first, as per investigator assessment and per blinded independent central review using RECIST v 1.1.
Overall survival (OS) | Baseline up to 24 months
  The time from randomization to death from any cause, as per investigator assessment and blinded independent central review using RECIST v 1.1.
Maximum tumor shrinkage (MTS) | Baseline up to 24 months
  The biggest decrease, or smallest increase if no decrease will be observed, as per investigator assessment and blinded independent central review using RECIST v 1.1.
Time to first subsequent therapy (TFST) | Baseline up to 24 months
  The time from randomization to the time a patient starts his/her first line treatment (first subsequent therapy).
Time to second subsequent therapy (TSST) | Baseline up to 24 months
  The time from randomization to the time a patient starts his/her second line treatment (second subsequent therapy).
Time to first chemotherapy (TFC) | Baseline up to 24 months
  The time from randomization to the time a patient included in Arm A starts his/her first line chemotherapy.
Incidence of adverse events (AEs) | Baseline up to 24 months
  Number of patients with treatment-related AEs (Grade 3 and 4 AEs and serious adverse events [SAEs]) by using the National Cancer Institute (NCI)-Common Terminology Criteria for Adverse Events (CTCAE) v.5.0.
Patient-reported global quality of life (QoL) | At the beginning of each cycle up to 36 months after study start.
  Overall change from baseline in patient-reported global QoL, general health status, functioning and symptoms; time to deterioration in global QoL; and time to deterioration in pain.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Llombart-Cussac, Principal Investigator — Arnau de Vilanova Hospital, Valencia (Spain)
Locations (31):
- Italy (4):
  - Instituto Europeo di Oncologia, Milan
  - Ospedale San Gerardo, Monza
  - Ospedale Guglielmo da Saliceto, Piacenza
  - Azienda Ospedaliero-Universitaria Cittá de la Salute e della Scienza, Torino
- Portugal (2):
  - Hospital Fernando da Fonseca, Amadora
  - Hospital de Santa Maria - Centro Hospitalar Lisboa Norte, Lisbon
- Spain (25):
  - Hospital Universitario Virgen del Rocio, Seville, Andalusia
  - Fundación Althaia Manresa, Manresa, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba, Cordoba
  - Centro Oncoloxico de Galicia, A Coruña, Coruña
  - Complejo Asistencial Universitario De León, León, Leon
  - Complejo Hospitalario de Navarra, Pamplona, Pamplona/Iruña
  - Hospital Universitari de Sant Joan de Reus, Reus, Tarragona
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Quiron Salud Dexeus, Barcelona
  - Hospital Universitario Basurto, Bilbao
  - Consorcio Hospitalario Provincial de Castellon, Castellon
  - Institut Catala D'Oncologia Girona - Hospital Josep Trueta, Girona
  - Hospital Universitario San Cecilio, Granada
  - Hospital Universitario Arnau de Vilanova, Lleida
  - Hospital Ruber Juan Bravo, Madrid
  - Hospital Beata María Ana, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario Clinico San Carlos, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Quirónsalud Sagrado Corazón, Seville
  - Hospital Clinico Universitario de Valencia, Valencia
  - Hospital Quironsalud Valencia, Valencia
  - Consorcio Hospital General Universitario de Valencia, Valencia
  - Hospital Arnau de Vilanova, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza

IPD SHARING:
Plan to Share IPD: No